CLINICAL TRIAL: NCT06904339
Title: Promoting Effective Clinical Communication About Sexual Health After Gynecologic Cancer: A Randomized Controlled Trial of a Patient-Focused Intervention
Brief Title: Communication About Sexual Health in Gynecologic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 24-1010; R01CA285674 (NIH)
Record Dates: First submitted 2025-03-31; First posted 2025-04-01 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Gynecologic Cancers
Keywords: sexual health

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sexual Health Resources Alone (Active Comparator): Participants will receive a resource guide with information on sexual health and gynecologic cancer. The guide will include organizational resources and links to websites with information about sexual health and gynecologic cancer.
  Interventions: Behavioral: Sexual Health Resources
- Sexual Health Resources + Starting the Conversation Video/Workbook (Experimental): Participants will receive a resource guide on sexual health and gynecologic cancer and will be asked to watch a 25-minute video with information about sexual health and gynecologic cancer and learn ways to talk to their cancer care provider effectively about sexual health concerns. Participants will also fill out a workbook with activities to help them practice communication skills and plan their discussion.
  Interventions: Behavioral: Starting the Conversation; Behavioral: Sexual Health Resources

INTERVENTIONS:
Behavioral: Starting the Conversation — Starting the Conversation includes a 25-minute video with information about sexual health and gynecologic cancer and tips about how to talk to their cancer care team about sexual health concerns. Participants will also fill out a workbook with activities to help them practice communication skills.
  Arms: Sexual Health Resources + Starting the Conversation Video/Workbook
Behavioral: Sexual Health Resources — The sexual health resource guide includes institutional resources for patients with sexual concerns (for example, the Women's Survivorship Clinic) and links to reputable websites with information about sexual health after gynecologic cancer.

SUMMARY:
The goal of this clinical trial is to learn if an educational video and workbook can help gynecologic cancer patients talk to their cancer providers about sexual health concerns.

The main questions it aims to answer are:

1. Do gynecologic cancer patients who take part in the educational program and get a resource booklet talk to their cancer clinicians more about sexual health concerns than patients who get a resource booklet alone?
2. Do gynecologic cancer patients who take part in the educational program and get a resource booklet have better sexual function and less anxiety and depression than patients who get a resource booklet alone?

Researchers will compare those who get the educational program and the resource booklet to those who get the resource booklet alone.

Participants will:

1. Fill out a consent form and survey
2. Have their next clinic visit audio recorded
3. Fill out another survey right after their clinic visit
4. Fill out a final survey 6 months after their clinic visit

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed with any stage (I-IV) gynecologic cancer
* Receiving treatment for gynecologic cancer or completed active treatment less than 10 years ago
* Attending visits in follow-up care at Fox Chase Cancer Center
* Score of at least 3 on a sexual concerns screener question

Exclusion Criteria:

* Not able to speak English
* Not willing to have clinic visit audio recorded
* Eastern Cooperative Oncology Group (ECOG) score > 2
* Overt cognitive dysfunction or psychiatric disturbance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Communication - Raise Topic of Sexual Health | 2 weeks
  Number of patients who raise the topic of sexual health concerns in a clinic visit.
Clinical Communication - Ask a Question about Sexual Health | 2 weeks
  Number of patients who ask a question about sexual health concerns in a clinic visit.
Clinical Communication - Express a Concern about Sexual Health | 2 weeks
  Number of patients who express a sexual health concern in a clinic visit.

SECONDARY OUTCOMES:
Self-Reported Sexual Function | Baseline, 2 weeks, 3 months, 6 months
  Patients' self-reported sexual function will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) SexFS Brief Profile Version 2.0. Four domains (lubrication, vaginal discomfort, satisfaction, and interest) will be scored. Domains are scored using T-scores, with higher scores signifying better sexual function for the lubrication, satisfaction, and interest domains. Lower scores in the vaginal discomfort range signify better sexual function.
Self-Reported Sexual Activity | Baseline, 2 weeks, 3 months, 6 months
  Patients' self-reported sexual activity will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sexual Activity screener. Number of participants reporting any sexual activity will be reported.
Self-Reported Anxiety Symptoms | Baseline, 2 weeks, 3 months, 6 months
  Patients' self-reported anxiety symptoms will be measured using the Hospital Anxiety and Depression Scale (HADS). The anxiety subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of anxiety.
Self-Reported Depressive Symptoms | Baseline, 2 weeks, 3 months, 6 months
  Patients' self-reported depressive symptoms will be measured using the Hospital Anxiety and Depression Scale (HADS). The depression subscale consists of 7 items that are scored from 0 to 3. Summed scores range from 0 to 21, with higher scores indicating higher levels of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No